CLINICAL TRIAL: NCT01677104
Title: The Microvascular Function of GLP-1 and Its Analogues in Humans, in Vivo: the Role of DPP-IV Inhibition
Brief Title: The Microvascular Function of GLP-1 and Its Analogues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Katarina Kos (Other)
Collaborators: Diabetes UK (Other)
Responsible Party: Sponsor-Investigator, Katarina Kos, Consultant Physician and Senior Lecturer, Royal Devon and Exeter NHS Foundation Trust
Organization: Royal Devon and Exeter NHS Foundation Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 11/SW/0195; 1204620 (Other: Research and Development)
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: GLP-1; DPP-IV inhibitor; microcirculation; Exenatide; Liraglutide; Linagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Glucagon-Like Peptide 1; Exenatide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DPP-IV inhibitor (Active Comparator): Linagliptin 5mg (Tradjenta) before microinjection of GLP-1 and its analogues
  Interventions: Drug: GLP-1; Drug: Placebo
- Placebo pill (Placebo Comparator): One placebo tablet before microinjection
  Interventions: Drug: GLP-1; Drug: Placebo

INTERVENTIONS:
Drug: GLP-1 — GLP-1 and its analogues will be compared with placebo with and without prior DPP-IV inhibition
  Other Names: native GLP-1(7,36); Exenatide (Byetta); Liraglutide (Vicotza)
Drug: Placebo

SUMMARY:
Incretins have become a successful drug target in the repertoire of medications used for the treatment of type 2 diabetes. However little is known about a potential benefit of GLP-1 on the vascular system in humans, independent of their glucose lowering actions and data are only derived from ex vivo studies in animals. Particularly little is known about clinically relevant benefits of GLP-1 and its analogues on the microvascular system of individuals with type 2 diabetes.

The vascular effect could be medicated by endogenous GLP-1 (9,36) amide, the breakdown product of GLP-1 (7,36) amide which has a low affinity for the GLP-1 receptor. The investigators hypothesis is that the co-administration of DPP-IV inhibitors will lack the beneficial effects of GLP-1 on the vascular system as GLP-1 (9,36) amide will not be produced by the body.

The study aims to examine the response of GLP-1 and its analogues on small blood vessels and examine the effect of the addition of DPP-IV inhibition in healthy lean individuals, obese individuals and subjects with Type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Lean BMI ≤ 25.0 kg/m2
* Obese BMI ≥30.0kg/m2
* Non diabetic subjects and subjects with Type 2 diabetes on stable medication for at least 3 months

Exclusion Criteria:

* cardiovascular disease
* Raynaud's disease
* current treatment with any anti-hypertensive
* lipid lowering therapies
* severe hepatic impairment
* pregnancy and lactation
* subjects with Type 2 diabetes on insulin therapy
* subjects with Type 2 diabetes on sulphonylureas
* subjects with Type 2 diabetes on incretin based therapies
* subjects with Type 2 diabetes and peripheral vascular disease
* subjects with Type 2 diabetes and history of advanced retinopathy
* subjects with Type 2 diabetes and advanced nephropathy
* subjects with Type 2 diabetes with uncontrolled diabetes (HbA1c > 8.5%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
skin blood flow | 3 hours
  skin blood flow will be assessed before and after microinjection of GLP-1 or its analogues and the injection site monitored and compared to sites injected with placebo

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Kos, MD, PHD, Principal Investigator — Institue of Biomedical and Clinical Sciences, Peninsula Medical School, University of Exeter
Locations (1):
- Diabetes and Vascular Center, Exeter, United Kingdom

REFERENCES:
- [Derived] Aung MM, Slade K, Freeman LAR, Kos K, Whatmore JL, Shore AC, Gooding KM. Locally delivered GLP-1 analogues liraglutide and exenatide enhance microvascular perfusion in individuals with and without type 2 diabetes. Diabetologia. 2019 Sep;62(9):1701-1711. doi: 10.1007/s00125-019-4918-x. Epub 2019 Jun 16. PMID 31203378